CLINICAL TRIAL: NCT03012620
Title: Secured Access to Pembrolizumab for Patients With Selected Rare Cancer Types
Acronym: AcSé
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1612; 2016-002260-14 (EudraCT Number)
Record Dates: First submitted 2017-01-02; First posted 2017-01-06 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Sarcoma; Ovarian Neoplasm; Central Nervous System Neoplasm; Thyroid Neoplasm; Carcinoma, Neuroendocrine; Neoplasms, Germ Cell and Embryonal; NK/T-cell Lymphoma
MeSH Terms: conditions — Sarcoma; Ovarian Neoplasms; Central Nervous System Neoplasms; Thyroid Neoplasms; Carcinoma, Neuroendocrine; Neoplasms, Germ Cell and Embryonal; Lymphoma, Extranodal NK-T-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg IV as a 30 minute infusion on Day 1 of every 21 day cycle
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Treatment
  Other Names: MK-3475; KEYTRUDA

SUMMARY:
This is a Phase 2, non-randomised, open-label, multicentric study to investigate the efficacy and safety of pembrolizumab monotherapy in 7 cohorts of patients with specific rare cancers who have unresectable locally advanced or metastatic disease, which is resistant or refractory to standard therapy, or for which standard therapy does not exist, or is not considered appropriate, and for which no other experimental treatment options are available, in order to identify subsets of patients that may benefit from treatment

DETAILED DESCRIPTION:
The study plans to enrol up to 350 patients in total. Eligible patients who have provided their written informed consent for study participation will be assigned to one of 7 cohorts determined by indication:

* Cohort 1: Rare sarcoma
* Cohort 2: Rare ovarian cancer
* Cohort 3: Primary central nervous system lymphomas
* Cohort 4: Rare thyroid cancer
* Cohort 5: Rare malignant neuroendocrine cancer
* Cohort 6: Germ-cell cancer
* Cohort 7: NK/T-cell lymphoma

Between 20 and 50 patients will be enrolled in each cohort with the exception of the cohort 1 for which up to 80 patients may be enrolled (extension introduced under amendment 5 of this protocol). Following the amendment 6, up to a maximum of 50 additional patients may be included in the Sarcoma (cohort 1), Rare ovarian cancer (cohort 2) or Primary central nervous system lymphoma (cohort 3) cohorts, within the limit of 350 patients to be included in total.

The study will use a two-stage Bayesian enrichment design. The first stage treats all patients from the different cohorts with the investigational product and identifies possibly sensitive indications. The second stage will compare outcomes among subsets of patients in the identified cohorts to distinguish between subpopulations of patients who may benefit from the treatment and patients for whom there is no evidence of efficacy.

All participants who reach the maximum treatment duration per protocol and stop the pembrolizumab with a clinical benefit (prolonged stable disease, partial or complete response), may be eligible for up to an additional 1 year (approximately 17 cycles) of pembrolizumab treatment if they progress during the follow-up period. This retreatment is termed the Second course or Re-challenge.

The second pembrolizumab course will continue until 12 months of retreatment, progression or until the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient information sheet and written informed consent form signed.
2. Histologically confirmed diagnosis of a pathology corresponding to one of the following selected cancer types:

   * Rare sarcoma: Alveolar soft part sarcoma, Chordoma, Dedifferentiated chondrosarcoma, epithelioid sarcoma, sarcoma with loss of INI1, malignant rhabdoid tumours, myxoid liposarcoma, angiosarcoma of the scalp, radiation induced sarcomas.From the 51st patient included in this cohort, only the following histological types will be selected: Alveolar soft part sarcoma, Chordoma, SMARCA4-malignant rhabdoid tumours and Desmoplastic small-round-cell tumor.
   * Rare ovarian cancer: recurrent or relapsed; sex cord tumour, germ cell tumour (immature teratoma, non seminomatous germ cell & dysgerminoma), low-grade serous carcinoma, mucinous carcinoma, clear cell adenocarcinoma, small cell carcinoma, and carcinosarcoma - with histological confirmation following review by members of the Tumeurs Malignes Rares Gynécologiques (TMRG) network (French rare gynaecological tumour group).From the 51st patient included in this cohort, only the following histological types will be selected: teratoma, low-grade serous carcinoma and ovarian small cell carcinoma hypercalcemic type (SCOOHT).
   * Primary central nervous system lymphoma (PCNSL): refractory primary intraocular and CNS lymphoma.From the 51st patient included in this cohort, only CNS lymphoma will be selected.
   * Rare thyroid cancer: differentiated thyroid carcinoma (Papillary, follicular, Hurthle cell (oncocytic), poorly differentiated thyroid carcinoma), medullary thyroid carcinoma, anaplastic thyroid carcinoma.
   * Rare malignant neuroendocrine tumour: poorly differentiated tumours refractory after 2 lines of chemotherapy, well differentiated tumours refractory after 4 lines of treatment, carcinoid tumours after 2 lines of treatment.
   * Germ-cell cancer progressing after standard therapy.
   * Natural killer T-cell lymphoma: extranodal NK/T-cell lymphoma regardless of localization that is resistant or refractory to prior L-asparaginase therapy.
3. Metastatic disease or unresectable locally advanced malignancy that is resistant or refractory to standard therapy or for which standard therapy does not exist or is not considered appropriate by the Investigator.
4. Aged ≥18 years old for cohort 2 to 7 and aged ≥15 years old for patients included in cohort 1 (rare sarcoma).
5. Measurable disease according to RECIST v1.1 guidelines for solid tumours; or International primary central nervous system lymphoma cooperative group (IPCG) response criteria for patients in the PCNSL cohort. For patients with germ-cell cancer measurable disease is defined as measurable according to RECIST v1.1 and / or abnormal levels of alpha-fetoprotein (AFP), human chorionic gonadotropin (hCG) and lactate dehydrogenase (LDH). For patients with NK/T-cell lymphoma measurable disease is defined as focal uptake in at least one nodal or extra-nodal site with a Lugano 5-PS score of 4 or 5.
6. Able to provide a Formalin-fixed/paraffin-embedded (FFPE) biopsy sample of a metastatic site or primitive tumour tissue.

   Note: Patients for whom suitable archived biopsy material is not available must be willing to undergo a biopsy of a tumour lesion prior to study entry, unless this is medically contraindicated (e.g. site inaccessible or patient safety concerns).
7. Patients must have a mandatory treatment-free interval of at least 21 days following previous systemic anti-cancer treatments.
8. Patients who have received previous systemic anticancer treatment and/or radiotherapy should have recovered from any treatment related toxicity, to a level of ≤ grade 1 (according to NCI-CTCAE criteria, v 4.0) with the exception of Grade 2 alopecia.
9. Adequate hematologic function (absolute neutrophil count (ANC) ≥1.0 x10⁹/L, platelets ≥100 x10⁹/L, haemoglobin ≥9 g/L) measured within 14 days of treatment initiation.
10. Adequate renal function (creatinine clearance ≥50 mL/min using the Modification of Diet in Renal Disease (MDRD) or CKI EPI method) measured within 14 days of treatment initiation.
11. Adequate hepatic function (serum bilirubin ≤1.5 x the reference upper limit of normal (ULN) unless due to Gilbert's syndrome; aspartate aminotransferase(ASAT) and alanine aminotransferase (ALAT) ≤2.5 x ULN) measured within 14 days of treatment initiation. For patients with documented liver metastasis ASAT/ALAT ≤ 5 x ULN is acceptable.
12. Strictly normal blood levels of calcium and magnesium, measured within 14 days of treatment initiation.
13. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤1.
14. Estimated life expectancy ≥90 days.
15. Patients who are sexually active must agree to use a medically accepted method of contraception (e.g. implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner, for participating women; condoms for participating men) or practice complete abstinence, beginning 14 days before the first administration of the investigational product (IP), while on treatment and for at least 5 months after the last administration of IP for female patients, and 7 months after the last administration of IP for male patients.
16. Women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to the first administration of IP. If urine test results are positive or cannot be confirmed as negative, a serum pregnancy test will be required.
17. Women who are breastfeeding should discontinue nursing prior to the first administration of IP and for at least 120 days after the last administration of IP.
18. Patients must be affiliated to a Social Security System or equivalent.

Exclusion Criteria:

1. Prior treatment with an anti-PD1 or anti-PD-L1 antibody
2. Eligible, and willing, to participate in a clinical trial of an alternative anticancer therapy targeting their disease which is open to accrual in France.
3. Concurrent steroid medication at a dose greater than prednisone 10 mg/day or equivalent. For patients with PCNSL or germ-cell cancer, concurrent steroid medication at a dose greater than prednisone 20 mg/day or equivalent.
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
5. History of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
6. History of severe hypersensitivity reaction to any monoclonal antibody therapy
7. Radiotherapy (except for brain and extremities) within 21 days prior to the first administration of IP.
8. Treatment with other investigational drugs or participation in another clinical trial within 21 days prior to the first administration of IP or concomitantly with the trial.
9. Has known symptomatic central nervous system (CNS) metastases. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
10. Has known carcinomatous meningitis or a history of leptomeningeal disease, except for patients with primary CNS lymphoma.
11. Serum creatinine >1.5 x ULN or glomerular filtration rate (GFR) <50 ml/min.
12. Other malignancies within the past 5 years other than basal cell skin cancer or in situ carcinoma of the cervix.
13. Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy.
14. Active or chronic hepatitis B, hepatitis C and/or human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies), or a known history of active Tuberculosis bacillus.
15. Has received a live vaccine within 30 days of planned start of study treatment. Note: Seasonal influenza vaccines for injection are generally inactivated vaccines and are allowed.
16. Active alcohol or drug abuse.
17. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule.
18. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Objective response rate | measured at the first scheduled disease assessment following study treatment initiation (Day 84, ± 7 days)
  ORR will be assessed per cohort by an IRC according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival | From date of inclusion until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Assessed according to RECIST v1.1
Overall survival | From date of inclusion until the date of death from any cause, assessed up to 36 months
Best response | From inclusion up to 36 months
  Assessed according to RECIST v1.1
Response duration | from first observation of objective response until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Assessed according to RECIST v1.1
Time to response | from inclusion first observation of objective response, assessed up to 36 months
  Assessed according to RECIST v1.1
Frequency and severity of adverse events | from inclusion until 100 days after last dose of investigational product
  Assessed according to the NCI-CTCAE v4
Objective response rate in subgroups of subjects with high versus low expression (cutoff set at the median for the population measured) of different immune markers (PD-L1, CD4+, FOXP3+, Fas-L, OX40, VEGF, CD31; CD34) | measured at the first scheduled disease assessment following study treatment initiation (Day 84, ± 7 days)
  ORR will be assessed per cohort by an IRC according to RECIST v1.1
Progression-free survival in subgroups of subjects with high versus low expression (cutoff set at the median for the population measured) of different immune markers (PD-L1, CD4+, FOXP3+, Fas-L, OX40, VEGF, CD31; CD34) | From date of inclusion until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Assessed according to RECIST v1.1
Overall survival in subgroups of subjects with high versus low expression (cutoff set at the median for the population measured) of different immune markers (PD-L1, CD4+, FOXP3+, Fas-L, OX40, VEGF, CD31; CD34) | From date of inclusion until the date of death from any cause, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Massard, MD, Principal Investigator — Gustave Roussy Cancer Campus
Locations (1):
- Gustave Roussy Cancer Campus, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blay JY, Chevret S, Le Cesne A, Brahmi M, Penel N, Cousin S, Bertucci F, Bompas E, Ryckewaert T, Soibinet P, Boudou-Rouquette P, Saada Bouzid E, Soulie P, Valentin T, Lotz JP, Tosi D, Neviere Z, Cancel M, Ray-Coquard I, Gambotti L, Legrand F, Lamrani-Ghaouti A, Simon C, Even C, Massard C. Pembrolizumab in patients with rare and ultra-rare sarcomas (AcSe Pembrolizumab): analysis of a subgroup from a non-randomised, open-label, phase 2, basket trial. Lancet Oncol. 2023 Aug;24(8):892-902. doi: 10.1016/S1470-2045(23)00282-6. Epub 2023 Jul 7. PMID 37429302